CLINICAL TRIAL: NCT00454649
Title: A Phase 1 Dose-Finding Study Of The Anti-Angiogenesis Agent, AG-013736, In Combinations Of Paclitaxel/Carboplatin, Weekly Paclitaxel, Docetaxel, Capecitabine, Gemcitabine/Cisplatin and Pemetrexed/Cisplatin In Patients With Advanced Solid Tumors
Brief Title: Investigational Agent AG-013736 In Combinations With Standard Of Care Treatments For Patient's With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061019
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Neoplasms
Keywords: axitinib; chemotherapy; anti-angiogenesis; VEGF inhibition
MeSH Terms: conditions — Neoplasms | interventions — Axitinib; Paclitaxel; Carboplatin; Docetaxel; Capecitabine; Gemcitabine; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axitinib [AG-013736] + chemotherapy combination (Experimental): The following separate groups were included:
  axitinib
  1. plus carboplatin/paclitaxel in three different schedules
  2. plus paclitaxel
  3. plus docetaxel/carboplatin
  4. plus docetaxel
  5. plus capecitabine
  6. plus gemcitabine/cisplatin
  7. plus pemetrexed/cisplatin
  Interventions: Drug: Axitinib + Paclitaxel + Carboplatin (Cohort 1); Drug: Axitinib + Paclitaxel + Carboplatin (Cohort 2); Drug: Axitinib + Paclitaxel + Carboplatin (Cohort 3); Drug: Axitinib + Paclitaxel (Cohort 4); Drug: Axitinib + Docetaxel + Carboplatin (Cohort 4a); Drug: Axitinib + Docetaxel (Cohort 5); Drug: Axitinib + Capecitabine (Cohort 6); Drug: Axitinib + Capecitabine (Cohort 7); Drug: Axitinib + Gemcitabine + Cisplatin (Cohort 8); Drug: Axitinib + Pemetrexed + Cisplatin (Cohort 9)

INTERVENTIONS:
Drug: Axitinib + Paclitaxel + Carboplatin (Cohort 1) — Axitinib (AG-013736) 1 milligram (mg) tablet orally twice daily (BID) as lead in dose from Day -5, -4 or -3 through Day 2 of Cycle 1 (21 days). Axitinib (AG-013736) 5 mg tablet orally BID from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 (21 days) and all subsequent cycles (21 days). Paclitaxel [200 milligram/square meter (mg/m^2)] 3-hour infusion followed by carboplatin 30-minutes infusion at a dose to target area under the concentration-time curve (AUC) of 6.0 milligram*minute/milliliter (mg*min/mL) on Day 1 of Cycle 1 and all subsequent cycles.
Drug: Axitinib + Paclitaxel + Carboplatin (Cohort 2) — Axitinib (AG-013736) 3 tablets of 1 mg orally BID as lead in dose from Day -5, -4 or -3 through Day 2 of Cycle 1 (21 days). Axitinib (AG-013736) 5 mg tablet orally BID from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 (21 days) and all subsequent cycles (21 days). Paclitaxel (200 mg/m^2) 3-hour infusion followed by carboplatin 30-minutes infusion at a dose to target AUC of 6.0 mg*min/mL on Day 1 of Cycle 1 and all subsequent cycles.
Drug: Axitinib + Paclitaxel + Carboplatin (Cohort 3) — Axitinib (AG-013736) 5 mg tablet orally BID as lead in dose from Day -5, -4 or -3 through Day 2 of Cycle 1 (21 days). Axitinib (AG-013736) 5 mg tablet orally BID from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 (21 days) and all subsequent cycles (21 days). Paclitaxel (200 mg/m^2) 3-hour infusion followed by carboplatin 30-minutes infusion at a dose to target AUC of 6.0 mg*min/mL on Day 1 of Cycle 1 and all subsequent cycles.
Drug: Axitinib + Paclitaxel (Cohort 4) — Axitinib (AG-013736) 5 mg tablet orally BID from Day 1 to Day 25 of Cycle 1 (28 days) and then without interruption from Day 3 for Cycle 2 (28 days) and all subsequent cycles (28 days). Paclitaxel (90 mg/m^2) 60-minute infusion on Day 1, 8, and 15 of each cycle.
Drug: Axitinib + Docetaxel + Carboplatin (Cohort 4a) — Axitinib (AG-013736) 5 mg tablet orally BID as lead in dose from Day -5, -4 or -3 through Day 2 of Cycle 1 (21 days). Axitinib (AG-013736) 5 mg tablet orally BID from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 (21 days) and all subsequent cycles (21 days). Docetaxel (75 mg/m^2) 60-minute infusion on Day 1 of every cycle. Carboplatin 30-minutes infusion at a dose to target AUC of 6.0 mg*min/mL on Day 1 of Cycle 1 and all subsequent cycles.
Drug: Axitinib + Docetaxel (Cohort 5) — Axitinib (AG-013736) 5 mg tablet orally BID as lead in dose from Day -5, -4 or -3 through Day 2 of Cycle 1. Axitinib (AG-013736) 5 mg oral tablet BID administered from Day 3 to Day 18 of Cycle 1 (21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles. Docetaxel (100 mg/m^2) 60-minute infusion on Day 1 of each cycle.
Drug: Axitinib + Capecitabine (Cohort 6) — Axitinib (AG-013736) 5 mg tablet orally BID from Day 1 to Day 18 of Cycle 1 (21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles. Capecitabine (1000 mg/m^2) orally BID from Day 1 to Day 14 of each cycle.
Drug: Axitinib + Capecitabine (Cohort 7) — Axitinib (AG-013736) 5 mg tablet orally BID from Day 1 to Day 18 of Cycle 1 (21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles. Capecitabine (1250 mg/m^2) orally BID from Day 1 to Day 14 of each cycle.
Drug: Axitinib + Gemcitabine + Cisplatin (Cohort 8) — Axitinib (AG-013736) 5 mg tablet orally BID from Day -5, -4 or -3 to Day 18 of Cycle 1 (21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles. Gemcitabine (1250 mg/m^2) 30-minute infusion on Day 1 and Day 8 of Cycle 1 and all subsequent cycles followed by cisplatin (80 mg/m^2) infusion on Day 1 of each cycle.
Drug: Axitinib + Pemetrexed + Cisplatin (Cohort 9) — Axitinib (AG-013736) 5 mg tablet orally BID from Day -5, -4 or -3 to Day 18 of Cycle 1 (21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles. Pemetrexed (500 mg/m^2) 10-minute infusion followed by cisplatin (75 mg/m^2) infusion on Day 1 of each cycle.

SUMMARY:
To determine the best dose of this investigational agent AG-013736 in combination with various standard of care treatments for advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors suitable for treatment with Taxanes, with or without carboplatin, or treatment with Capecitabine, Gemcitabine/Cisplatin. or Pemetrexed/Cisplatin

Exclusion Criteria:

* Tumors abutting or providing support for blood vessels
* Any significant gastrointestinal abnormalities or active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-12; Primary Completion 2009-08 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (8):
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Harvey, Illinois
  - Pfizer Investigational Site, Tinley Park, Illinois
  - Pfizer Investigational Site, Hobart, Indiana
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Kennewick, Washington
- Pfizer Investigational Site, Warsaw, Poland
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061019&StudyName=Investigational%20Agent%20AG-013736%20In%20Combinations%20With%20Standard%20Of%20Care%20Treatments%20For%20Patient%27s%20With%20Advanced%20Solid%20Tumor

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 102 participants were enrolled for the study. Out of those, 4 participants were screen failure and were not included in results analysis.
Period: Overall Study
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel + Carboplatin (Cohort 4a) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Started | 3 | 5 | 20 | 7 | 1 | 7 | 9 | 19 | 21 | 6
Completed | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not Completed | 3 | 4 | 19 | 6 | 1 | 7 | 9 | 19 | 20 | 5
Not completed — Lack of Efficacy | 2 | 2 | 10 | 3 | 0 | 4 | 5 | 13 | 10 | 2
Not completed — Adverse Event | 0 | 1 | 3 | 0 | 1 | 2 | 3 | 4 | 6 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 5 | 3 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel + Carboplatin (Cohort 4a) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9) | Total
Number analyzed (Participants) | 3 | 5 | 20 | 7 | 1 | 7 | 9 | 19 | 21 | 6 | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (11.4) | 62 (16.6) | 59.5 (10.6) | 60.7 (10.2) | 64 (NA) — Standard deviation was not calculated as only one participant was evaluable. | 63.4 (11.9) | 60.4 (12.4) | 53.4 (10.6) | 54 (10.3) | 58.8 (9.0) | 57.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 3 | 1 | 5 | 5 | 11 | 12 | 3 | 47
  Male | 1 | 3 | 17 | 4 | 0 | 2 | 4 | 8 | 9 | 3 | 51

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Axitinib (AG-013736) in Combination With Chemotherapy
Description: MTD defined as the dose level at which more than 1 out of 6 participants experienced a dose limiting toxicity (DLT). DLT included grade (Gr) 4 neutropenia or thrombocytopenia, greater than or equal to (>=) Gr 3 nonhematological toxicities or >=0.5 teaspoon/day hemoptysis or >=2 gram /24 hours proteinuria or inability to resume background chemotherapy or axitinib (AG-013736) dosing within 14 days of stopping due to treatment related toxicity.
Time Frame: Baseline to withdrawal from study or Day 21 of Cycle 1 [all cohorts except cohort 4 (Day 28 of Cycle 1)]
Population: Safety analysis population included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg BID
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 3 | 5 | 20 | 7 | 7 | 9 | 19 | 21 | 6
mg BID | 5 | 5 | 5 | 5 | NA — Axitinib (AG-013736) 5 mg BID was determined to be above the MTD. | 5 | 5 | 5 | 5

2. Secondary Outcome: Area Under the Curve From Time Zero to Time 24 Hours [AUC (0-24)] for Axitinib (AG-013736)
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero (pre-dose) to time 24 hours (0-24).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 hr post-dose on Day -1 for cohort 1, 2, 3, 5 and 8; on Day 22 of Cycle 1 for cohort 4; on Day 18 of Cycle 1 for cohorts 6 and 7; 0 (pre-dose), 1.2, 2.2, 3.2, 4.2, 6.2, 8.2 hr post-dose on Day -1 for cohort 9
Population: The pharmacokinetic parameter analysis set included all treated participants who had at least 1 estimated pharmacokinetic parameter of primary interest. N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- Axitinib + Paclitaxel + Carboplatin (Cohort 1): Axitinib (AG-013736) oral tablet of 1 mg (milligram) administered twice daily (BID) as lead in dose from Day -5, -4 or -3 to Day 2 of Cycle 1 (cycle length 21 days). AG-013736 standard dose of 5 mg oral tablet BID administered from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 and all subsequent cycles with no interval between two cycles. Paclitaxel [200 milligram/square meter (mg/m^2)] 3-hour infusion followed by carboplatin at a dose to target area under the concentration-time curve (AUC) of 6.0 milligram*minute/milliliter (mg*min/mL) as 30-minute infusion administered once weekly from Day 1 of Cycle 1 and all subsequent cycles.
- Axitinib + Paclitaxel + Carboplatin (Cohort 2): AG-013736 3 oral tablets of 1 mg administered BID as lead in dose from Day -5, -4 or -3 to Day 2 of Cycle 1 (cycle length 21 days). AG-013736 standard dose of 5 mg oral tablet BID administered from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 and all subsequent cycles with no interval between two cycles. Paclitaxel (200 mg/m^2) 3-hour infusion followed by carboplatin at a dose to target AUC of 6.0 mg*min/mL as 30-minute infusion administered once weekly from Day 1 of Cycle 1 and all subsequent cycles.
- Axitinib + Paclitaxel + Carboplatin (Cohort 3): AG-013736 oral tablet of 5 mg administered BID as lead in dose from Day -5, -4 or -3 to Day 2 of Cycle 1 (cycle length 21 days). AG-013736 standard dose of 5 mg oral tablet BID administered from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 and all subsequent cycles with no interval between two cycles. Paclitaxel (200 mg/m^2) 3-hour infusion followed by carboplatin at a dose to target AUC of 6.0 mg*min/mL as 30-minute infusion administered once weekly from Day 1 of Cycle 1 and all subsequent cycles.
- Axitinib + Paclitaxel (Cohort 4): AG-013736 oral tablet of 5 mg administered BID from Day 1 to Day 25 of Cycle 1 (cycle length 28 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles with no interval between two cycles. Paclitaxel 90 mg/m^2 administered as 60-minute infusion on Day 1, 8, and 15 of every cycle.
- Axitinib + Docetaxel (Cohort 5): AG-013736 oral tablet of 5 mg administered BID as lead in dose from Day -5, -4 or -3 to Day 2 of Cycle 1. AG-013736 standard dose of 5 mg oral tablet BID administered from Day 3 to Day 18 of Cycle 1 (cycle length 21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles with no interval between two cycles. Docetaxel 100 mg/m^2 administered as 60-minute infusion on Day 1 of every cycle.
- Axitinib + Capecitabine (Cohort 6): AG-013736 oral tablet of 5 mg administered BID from Day 1 to Day 18 of Cycle 1 (cycle length 21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles with no interval between two cycles. Capecitabine (1000 mg/m^2) administered orally BID from Day 1 to Day 14 of every cycle.
- Axitinib + Capecitabine (Cohort 7): AG-013736 oral tablet of 5 mg administered BID from Day 1 to Day 18 of Cycle 1 (cycle length 21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles with no interval between two cycles. Capecitabine (1250 mg/m^2) administered orally BID from Day 1 to Day 14 of every cycle.
- Axitinib + Gemcitabine + Cisplatin (Cohort 8): AG-013736 oral tablet of 5 mg administered BID from Day -5, -4 or -3 to Day 18 of Cycle 1 (cycle length 21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles with no interval. Cisplatin 80 mg/m^2 administered as infusion on Day 1 of Cycle 1 and all subsequent cycles. Gemcitabine 1250 mg/m^2 administered as infusion on Day 1 and Day 8 of Cycle 1 and all subsequent cycles.
- Axitinib + Pemetrexed + Cisplatin (Cohort 9): AG-013736 oral tablet of 5 mg administered BID from Day -5, -4 or -3 to Day 18 of Cycle 1 (cycle length 21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles with no interval between two cycles. Cisplatin 75 mg/m^2 and pemetrexed 500 mg/m^2 administered as infusion on Day 1 Cycle 1 and all subsequent cycles.
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 3 | 5 | 4 | 3 | 6 | 6 | 9 | 15 | 3
nanogram*hour/milliliter (ng*hr/mL) | 61.58 (54.66) | 242.41 (132.24) | 475.18 (380.13) | 154.43 (28.93) | 780.99 (535.30) | 365.95 (143.13) | 449.99 (323.59) | 416.30 (450.43) | 420.64 (200.32)

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Axitinib (AG-013736)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 3 | 5 | 6 | 5 | 7 | 7 | 15 | 20 | 4
ng/mL | 5.97 (2.59) | 23.36 (8.08) | 42.58 (18.25) | 44.58 (44.78) | 67.96 (39.24) | 37.51 (15.31) | 43.97 (28.82) | 40.97 (33.06) | 31.53 (22.87)

4. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Axitinib (AG-013736)
Time Frame: as for outcome 2
Population: Data was not summarized as majority of participants were having plasma concentrations below limit of assay quantification (BLQ).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Apparent Oral Clearance (CL/F) for Axitinib (AG-013736)
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes and F is the absolute oral bioavailability. Apparent oral clearance(CL/F) is obtained following oral administration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hour (L/hr)
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 3 | 5 | 4 | 3 | 6 | 6 | 9 | 15 | 3
Liter/hour (L/hr) | 49.39 (34.46) | 40.72 (46.75) | 29.73 (18.49) | 65.69 (11.94) | 14.35 (7.67) | 26.64 (15.58) | 83.46 (171.05) | 50.05 (56.75) | 25.10 (21.31)

6. Secondary Outcome: Plasma Decay Half Life (t1/2) for Axitinib (AG-013736)
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 3 | 5 | 4 | 3 | 6 | 6 | 9 | 15 | 3
hr | 2.75 (2.06) | 2.90 (1.78) | 2.80 (1.04) | 1.45 (0.27) | 4.07 (2.60) | 3.85 (1.93) | 3.64 (2.03) | 2.68 (1.09) | 5.02 (3.38)

7. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)] for Paclitaxel
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (pre-dose), 1, 2, 3, 3.25, 3.5, 4, 5, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 1-3; 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3): Combined Data from all participants in cohort 1, 2 and 3.
Arm/Group | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 6 | 12
ng*hr/mL | 5683.55 (1519.49) | 19959.91 (5951.86)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Paclitaxel
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 6 | 12
ng/mL | 3698.33 (1198.32) | 6105.00 (2167.59)

9. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Paclitaxel
Time Frame: as for outcome 7
Population: Cmin was analyzed only for orally administered drugs.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Plasma Clearance (CL) for Paclitaxel
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the plasma.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 6 | 12
L/hr | 30.48 (6.16) | 21.61 (9.38)

11. Secondary Outcome: Plasma Decay Half Life (t1/2) for Paclitaxel
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 6 | 12
hr | 12.51 (1.03) | 8.36 (2.16)

12. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)] for Docetaxel
Description: as for outcome 7
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Docetaxel (Cohort 5)
Number analyzed (Participants) | 4
ng*hr/mL | 3478.49 (870.12)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Docetaxel
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Docetaxel (Cohort 5)
Number analyzed (Participants) | 5
ng/mL | 3130.00 (1106.23)

14. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Docetaxel
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 5
Population: Cmin was analyzed only for orally administered drugs.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Docetaxel (Cohort 5)
Number analyzed (Participants) | 0

15. Secondary Outcome: Plasma Clearance (CL) for Docetaxel
Description: as for outcome 10
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Axitinib + Docetaxel (Cohort 5)
Number analyzed (Participants) | 4
L/hr | 42.96 (6.04)

16. Secondary Outcome: Plasma Decay Half Life (t1/2) for Docetaxel
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 24, 30 hr after start of infusion on Day 1 of Cycle 2 for cohort 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Docetaxel (Cohort 5)
Number analyzed (Participants) | 4
hr | 11.49 (0.97)

17. Secondary Outcome: Area Under the Curve From Time Zero to Time 24 Hours [AUC (0-24)] for Capecitabine
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero (pre-dose) to time 24 hours (0-24).
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hr post-dose on Day 1 of Cycle 2 for cohort 6 and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7)
Number analyzed (Participants) | 3 | 13
ng*hr/mL | 20534.52 (3797.63) | 22163.88 (16881.96)

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Capecitabine
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hr post-dose on Day 1 of Cycle 2 for cohort 6 and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7)
Number analyzed (Participants) | 5 | 16
ng/mL | 10808.00 (6173.62) | 10588.38 (9954.76)

19. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Capecitabine
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hr post-dose on Day 1 of Cycle 2 for cohort 6 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Apparent Oral Clearance (CL/F) for Capecitabine
Description: as for outcome 5
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hr post-dose on Day 1 of Cycle 2 for cohort 6 and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/hr
Arm/Group | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7)
Number analyzed (Participants) | 3 | 13
Liter/hr | 209.05 (24.29) | 314.12 (247.27)

21. Secondary Outcome: Plasma Decay Half Life (t1/2) for Capecitabine
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hr post-dose on Day 1 of Cycle 2 for cohort 6 and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7)
Number analyzed (Participants) | 3 | 13
hr | 0.85 (0.90) | 1.44 (3.05)

22. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)] for Gemcitabine
Description: as for outcome 7
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4 hr after start of infusion on Day 1 of Cycle 2 for cohort 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8)
Number analyzed (Participants) | 17
ng*hr/mL | 10991.16 (3099.28)

23. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Gemcitabine
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4 hr after start of infusion on Day 1 of Cycle 2 for cohort 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8)
Number analyzed (Participants) | 17
ng/mL | 20635.29 (10656.86)

24. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Gemcitabine
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4 hr after start of infusion on Day 1 of Cycle 2 for cohort 8
Population: Cmin was analyzed only for orally administered drugs.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8)
Number analyzed (Participants) | 0

25. Secondary Outcome: Plasma Clearance (CL) for Gemcitabine
Description: as for outcome 10
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4 hr after start of infusion on Day 1 of Cycle 2 for cohort 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8)
Number analyzed (Participants) | 17
L/hr | 224.36 (74.45)

26. Secondary Outcome: Plasma Decay Half Life (t1/2) for Gemcitabine
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4 hr after start of infusion on Day 1 of Cycle 2 for cohort 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8)
Number analyzed (Participants) | 17
hr | 0.29 (0.07)

27. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)] for Carboplatin
Description: as for outcome 7
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 5 hr after start of infusion on Day 1 of Cycle 2 for cohort 1-3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 12
ng*hr/mL | 55580.26 (9689.44)

28. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Carboplatin
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 5 hr after start of infusion on Day 1 of Cycle 2 for cohort 1-3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 12
ng/mL | 23383.33 (7170.75)

29. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Carboplatin
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 5 hr after start of infusion on Day 1 of Cycle 2 for cohort 1-3
Population: Cmin was analyzed only for orally administered drugs.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 0

30. Secondary Outcome: Plasma Clearance (CL) for Carboplatin
Description: as for outcome 10
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 5 hr after start of infusion on Day 1 of Cycle 2 for cohort 1-3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 12
L/hr | 12.57 (3.99)

31. Secondary Outcome: Plasma Decay Half Life (t1/2) for Carboplatin
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 5 hr after start of infusion on Day 1 of Cycle 2 for cohort 1-3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Combined Cohort 1, 2, 3)
Number analyzed (Participants) | 12
hr | 2.62 (0.55)

32. Secondary Outcome: Area Under the Curve From Time Zero to Time 8 Hours [AUC (0-8)] for Cisplatin
Description: AUC (0-8) = Area under the plasma concentration versus time curve from time zero (pre-dose) to time 8 hours (0-8).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 7 hr after start of infusion on Day 1 of Cycle 2 for cohort 8 and 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 12 | 4
ng*hr/mL | 2932.43 (929.69) | 2703.92 (688.68)

33. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Cisplatin
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 7 hr after start of infusion on Day 1 of Cycle 2 for cohort 8 and 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 13 | 4
ng/mL | 1680.54 (628.63) | 1176.00 (295.29)

34. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Cisplatin
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 7 hr after start of infusion on Day 1 of Cycle 2 for cohort 8 and 9
Population: Cmin was analyzed only for orally administered drugs.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Plasma Clearance (CL) for Cisplatin
Description: as for outcome 10
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 7 hr after start of infusion on Day 1 of Cycle 2 for cohort 8 and 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 12 | 4
L/hr | 46.31 (14.57) | 46.80 (14.92)

36. Secondary Outcome: Plasma Decay Half Life (t1/2) for Cisplatin
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 7 hr after start of infusion on Day 1 of Cycle 2 for cohort 8 and 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 12 | 4
hr | 2.61 (1.27) | 3.91 (1.59)

37. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)] for Pemetrexed
Description: as for outcome 7
Time Frame: 0 (pre-dose), 10 minutes (end of infusion), 0.5, 1, 1.5, 2, 4, 6, 8 hr after end of infusion on Day 1 of Cycle 2 for cohort 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 4
ng*hr/mL | 133032.97 (40176.65)

38. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Pemetrexed
Time Frame: as for outcome 37
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 4
ng/mL | 83925.00 (35820.05)

39. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Pemetrexed
Time Frame: as for outcome 37
Population: Cmin was analyzed only for orally administered drugs.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 0

40. Secondary Outcome: Plasma Clearance (CL) for Pemetrexed
Description: as for outcome 10
Time Frame: as for outcome 37
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 4
L/hr | 7.26 (2.08)

41. Secondary Outcome: Plasma Decay Half Life (t1/2) for Pemetrexed
Description: t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 37
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 4
hr | 2.77 (1.80)

42. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. Confirmed response are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline and thereafter every 2 cycles up to disease progression or discontinuation from study or up to 155 weeks
Population: Population included all participants who received at least 1 dose of study medication and had at least 1 target lesion according to RECIST and a baseline assessment of disease.
Measure: Number; unit: Percentage of Participants
Groups:
- Axitinib + Paclitaxel + Carboplatin (Cohort 1): Axitinib (AG-013736) 1 milligram (mg) tablet orally twice daily (BID) as lead in dose from Day -5, -4 or -3 through Day 2 of Cycle 1 (21 days). Axitinib (AG-013736) 5 mg tablet orally BID from Day 3 to Day 18 of Cycle 1 and Day 3 to Day 20 of Cycle 2 (21 days) and all subsequent cycles (21 days). Paclitaxel [200 milligram/meter square (mg/m^2)] 3-hour infusion followed by carboplatin 30-minutes infusion at a dose to target area under the concentration-time curve (AUC) of 6.0 milligram*minute/milliliter (mg*min/mL) on Day 1 of Cycle 1 and all subsequent cycles.
- Axitinib + Gemcitabine + Cisplatin (Cohort 8): Axitinib (AG-013736) 5 mg tablet orally BID from Day -5, -4 or -3 to Day 18 of Cycle 1 (21 days) and then without interruption from Day 3 of Cycle 2 and all subsequent cycles. Gemcitabine (1250 mg/m^2) 30-minute infusion on Day 1 and Day 18 of Cycle 1 and all subsequent cycles followed by cisplatin (80 mg/m^2) infusion on Day 1 of each cycle.
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Number analyzed (Participants) | 3 | 4 | 20 | 6 | 6 | 9 | 17 | 21 | 5
Percentage of Participants | 100.0 | 0 | 35.0 | 66.7 | 50.0 | 11.1 | 11.8 | 23.8 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib + Paclitaxel + Carboplatin (Cohort 1) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) | Axitinib + Paclitaxel (Cohort 4) | Axitinib + Docetaxel + Carboplatin (Cohort 4a) | Axitinib + Docetaxel (Cohort 5) | Axitinib + Capecitabine (Cohort 6) | Axitinib + Capecitabine (Cohort 7) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) | Axitinib + Pemetrexed + Cisplatin (Cohort 9)
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/5 | 11/20 | 2/7 | 1/1 | 4/7 | 6/9 | 9/19 | 13/21 | 4/6
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 20/20 | 7/7 | 1/1 | 7/7 | 9/9 | 19/19 | 21/21 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Paclitaxel + Carboplatin (Cohort 1) (N=3) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) (N=5) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) (N=20) | Axitinib + Paclitaxel (Cohort 4) (N=7) | Axitinib + Docetaxel + Carboplatin (Cohort 4a) (N=1) | Axitinib + Docetaxel (Cohort 5) (N=7) | Axitinib + Capecitabine (Cohort 6) (N=9) | Axitinib + Capecitabine (Cohort 7) (N=19) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) (N=21) | Axitinib + Pemetrexed + Cisplatin (Cohort 9) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Drug interaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1
Hypotension (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Paclitaxel + Carboplatin (Cohort 1) (N=3) | Axitinib + Paclitaxel + Carboplatin (Cohort 2) (N=5) | Axitinib + Paclitaxel + Carboplatin (Cohort 3) (N=20) | Axitinib + Paclitaxel (Cohort 4) (N=7) | Axitinib + Docetaxel + Carboplatin (Cohort 4a) (N=1) | Axitinib + Docetaxel (Cohort 5) (N=7) | Axitinib + Capecitabine (Cohort 6) (N=9) | Axitinib + Capecitabine (Cohort 7) (N=19) | Axitinib + Gemcitabine + Cisplatin (Cohort 8) (N=21) | Axitinib + Pemetrexed + Cisplatin (Cohort 9) (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 5 | 0 | 0 | 2 | 1 | 3 | 10 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 7 | 1 | 0 | 2 | 2 | 2 | 11 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 5 | 0 | 0 | 1 | 0 | 0 | 8 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Thyroid disorder (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1 | 3 | 3 | 3 | 6 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 3 | 4 | 0 | 3 | 2 | 2 | 11 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 7 | 5 | 1 | 4 | 4 | 14 | 8 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 0 | 3 | 0 | 1 | 4 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 0 | 1 | 0 | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 5 | 5 | 0 | 4 | 5 | 12 | 15 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 1 | 5 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 0 | 2 | 4 | 10 | 12 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 2 | 2 | 3 | 0 | 1 | 0 | 2 | 1 | 2 | 1
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 5 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 3 | 4 | 9 | 7 | 0 | 5 | 7 | 13 | 16 | 2
General physical health deterioration (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 5 | 4 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 3 | 1 | 0 | 1 | 1 | 2 | 3 | 0
Therapeutic response unexpected (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visceral oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 7 | 5 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Bacteria urine identified (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1
Blood culture positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eosinophils urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibrin D dimer (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 5 | 0 | 0 | 3 | 3 | 4 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 9 | 3 | 1 | 3 | 3 | 11 | 11 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2 | 0 | 4 | 4 | 2 | 8 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 0 | 2 | 1 | 4 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7 | 2 | 0 | 2 | 1 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 2 | 1 | 1 | 1 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 3 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 2 | 1 | 1 | 2 | 4 | 6 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 2 | 4 | 4 | 1 | 3 | 0 | 2 | 3 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 5 | 4 | 0 | 1 | 4 | 8 | 11 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 4 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 2 | 4 | 3 | 0 | 2 | 0 | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 5 | 1 | 0 | 1 | 0 | 4 | 2 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 2 | 3 | 1 | 0 | 2 | 0 | 4 | 6 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 7 | 2 | 0 | 2 | 1 | 3 | 5 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2 | 0 | 1 | 1 | 0 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 4 | 1 | 0 | 3 | 6 | 8 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 4 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal blistering (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4 | 9 | 4 | 1 | 4 | 0 | 0 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2 | 5 | 5 | 1 | 2 | 3 | 10 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 7 | 5 | 0 | 2 | 1 | 4 | 8 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 3 | 3 | 5 | 3 | 0 | 2 | 1 | 10 | 9 | 1
Hypotension (Vascular disorders) | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.